CLINICAL TRIAL: NCT00916240
Title: Multisystemic Therapy to Reduce Health Disparities in Adolescents With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sylvie Naar-King, PhD, Principal Investigator, Wayne State University School of Medicine, Department of Pediatrics
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 648; 1R01HL087272-01A1 (NIH)
Record Dates: First submitted 2009-06-05; First posted 2009-06-09 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2009-07

CONDITIONS: Asthma
Keywords: Adolescents; African American
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive Multisystemic Therapy (MST).
  Interventions: Behavioral: Multisystemic Therapy
- 2 (Active Comparator): Participants will receive home-based, non-directive family support.
  Interventions: Behavioral: Home-based, Non-Directive Family Support

INTERVENTIONS:
Behavioral: Multisystemic Therapy — Treatment will consist of a home- and community-based intensive intervention. Psychological treatment sessions will be provided in participants' homes, at a time designated by the participant and will last about 1 hour.
  Other Names: MST
  Arms: 1
Behavioral: Home-based, Non-Directive Family Support — Treatment will consist of Rogerian, client-centered, non-directive counseling. Participants will receive weekly home-based, supportive family counseling, with sessions lasting about 45 minutes.
  Arms: 2

SUMMARY:
Asthma is a chronic lung disease that inflames and narrows the airways. Symptoms can include recurring periods of wheezing, chest tightness, shortness of breath, and coughing. Minority, inner city teens are at increased risk for complications from the disease, possibly because of poor illness management. The purpose of this study is to test the effectiveness of Multisystemic Therapy (MST)-an intensive, home- and community-based psychotherapy-for improving asthma management and overall health and for reducing healthcare costs for inner city African American teens with asthma.

DETAILED DESCRIPTION:
Although rates of childhood asthma are increasing worldwide, more alarming is the disproportionate rise in rates of asthma among urban, disadvantaged, minority children. Inner city children, particularly adolescents, also appear to be most at risk for morbidity, mortality, and emergency department visits as a result of asthma. This may be caused by poor illness management.

Because of the multiple factors that affect whether or not a family is able to adequately manage a youth's asthma, educational interventions alone are typically insufficient to reduce morbidity and healthcare utilization, particularly in high-risk urban populations. As a result, more intensive, multi-component interventions are necessary to improve asthma management and outcomes for those youth at highest risk. MST is an innovative, flexible, home- and community-based family therapy that has been shown to improve health outcomes in urban children and adolescents with other chronic medical conditions such as type 1 diabetes and HIV infection. The purpose of this study is to determine the effectiveness of MST in improving health outcomes and reducing healthcare costs in high-risk urban adolescents with moderate to severe persistent asthma.

Participants will include high-risk African-American adolescents with moderate to severe asthma. High-risk youth are defined as those with one or more hospitalizations for asthma treatment in the previous 12 months. At a baseline hospital visit, participants will complete questionnaires and an interview, both of which will focus on the participant's family and asthma history. Participants will also have the option of having the study personnel visit their home instead. Participants will then be randomly assigned to receive either MST plus standard multidisciplinary specialty care or standard multidisciplinary care alone.

Participants assigned to MST will attend psychological treatment sessions in their homes for about 6 months. Treatment sessions will be attended by both children and parents, occur at a time designated by the participants, and last about 1 hour. Participants will also complete questionnaires about their interactions with the therapist and their satisfaction with treatment.

Participants assigned to standard multidisciplinary specialty care alone will receive weekly home-based, supportive family counseling for about 6 months. The treatment will provide emotional support to the family regarding asthma, help the family spot problems in asthma care, and address specific support that may help them with asthma management. Counseling sessions will last about 45 minutes.

Participants in both groups will receive treatment for 6 months and follow-up for 12 months. Participants will be evaluated at baseline and after 7 and 12 months. Families will also be contacted during Months 3 and 9 for medical information. During the study, the medical charts of participants with asthma will be reviewed for medical history and clinic visits. Other medical providers who directly care for the participant's asthma (e.g., primary care provider) may also be contacted. At the Month 6 evaluation, height and weight measurements will be taken.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe persistent asthma
* African American
* One or more hospitalizations for asthma in the last 12 months

Exclusion Criteria:

* No exclusions will be made due to co-morbid mental health problems (i.e., attention deficit hyperactivity disorder [ADHD], conduct disorder, depression, anxiety disorder), with the exception of thought disorder (i.e. schizophrenia, autism), suicidality, or mental retardation

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2008-09; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pulmonary functioning (FEV-1, FVC) | Measured at study entry and Months 7 (post treatment) and 12
Hospital and emergency department utilization (for asthma exacerbation) | Measured at study entry and Months 7 (post treatment) and 12

SECONDARY OUTCOMES:
Identification of mediators and moderators of MST treatment effects, e.g., individual adolescent factors (asthma knowledge/skill, mental health); family factors (family routines and relationships), etc. | Measured at study entry and Months 7 (post treatment) and 12

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Naar-King, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne State University School of Medicine, Detroit, Michigan, United States

REFERENCES:
- [Derived] Naar S, Ellis D, Cunningham P, Pennar AL, Lam P, Brownstein NC, Bruzzese JM. Comprehensive Community-Based Intervention and Asthma Outcomes in African American Adolescents. Pediatrics. 2018 Oct;142(4):e20173737. doi: 10.1542/peds.2017-3737. Epub 2018 Sep 5. PMID 30185428